CLINICAL TRIAL: NCT02192502
Title: A Randomized Controlled Investigation of the Effects of 6% Hydroxyethylstarch 130/0.4 (Voluven) on Renal Function in Patients Having Aortic Valve Replacement With or Without Coronary Artery Bypass Grafting
Brief Title: Use of 6% Hydroxyethylstarch (130/0.4) in Cardiac Surgical Patients
Acronym: SHARP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 012-973
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Kidney Injury
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HES 130/0.4 (Voluven) (Experimental): 6% HES 130/0.4 during surgery
  Interventions: Drug: HES 130/0.4 (Voluven)
- human albumin 5% (Active Comparator): human albumin 5% during surgery
  Interventions: Drug: human albumin 5%

INTERVENTIONS:
Drug: human albumin 5%
  Arms: human albumin 5%
Drug: HES 130/0.4 (Voluven)
  Arms: HES 130/0.4 (Voluven)

SUMMARY:
The purpose of this study is to evaluate the safety of a standard volume replacement called HES 130/0.4 (Voluven) during surgery on recovery. HES 130/0.4 (Voluven) may offer an alternative to pure fluid replacement solutions that are associated with problems after surgery including fluid overload and respiratory difficulties. The safety of HES 130/0.4 (Voluven) will be evaluated by examining its effects on kidney function, and coagulation parameters and platelet (part of the blood that help it clot) function.

Participants will be randomized (like flipping a coin) to receive one of two possible volume replacements during surgery, if fluid volume decreases enough to need replacement with one of the fluids. The two possible volume replacements are Voluven (a starch-containing fluid) or human albumin 5% (a protein-containing solution).

To examine kidney function, urine will be-sampled when the participant is put under general anesthesia, before surgical incision, within one hour of arrival to the ICU and 24 hours after completion of surgery. Two tubes (2 teaspoons) of blood (from an already established line) will be taken the morning of the surgery, within one hour of arrival to the ICU, 24 hours after surgery and every morning during the participants postoperative ICU stay.

Additionally, health and recovery information will be recorded from the participant's medical record. We will phone participants around 90 days and one year after surgery to ask a few questions about one's health and recovery. We will also record blood sample analysis results from follow up appointments within the first year after surgery. If this analysis is not conducted at the Cleveland Clinic, with permission, we will obtain the results from a treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 85 years old
* Scheduled for elective aortic valve replacement with or without coronary artery bypass grafting with or without additional minor surgical procedure.
* Written, informed consent for participation in this investigation.

Exclusion Criteria:

* Patients with renal failure with oliguria or anuria not related to hypovolemia.
* Patients receiving dialysis.
* Patients with preoperative renal insufficiency (Creatinine > 1.6 mg/dL)
* Anticipated deep hypothermic circulatory arrest
* Known hypersensitivity or allergy to hydroxyethyl starch or the excipients of hydroxyethyl starch
* Clinical conditions with volume overload (e.g., patients in pulmonary edema or congestive heart failure)
* Patients with severe hypernatremia or severe hyperchloremia
* Patients with intracranial bleeding
* Pregnant or breast feeding women
* Critically ill adult patients, including patients with sepsis, due to increased risk of mortality and renal replacement therapy, (e.g. patients who are hospitalized in the intensive care unit prior to surgery)
* Severe liver disease
* Pre-existing coagulation or bleeding disorders
* Any contraindications to proposed interventions.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andra Duncan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Lee MJ, Tannenbaum C, Mao G, Jia Y, Leung S, Yilmaz HO, Ince I, Soltesz E, Duncan AE. Effect of 6% Hydroxyethyl Starch 130/0.4 on Inflammatory Response and Pulmonary Function in Patients Having Cardiac Surgery: A Randomized Clinical Trial. Anesth Analg. 2021 Oct 1;133(4):906-914. doi: 10.1213/ANE.0000000000005664. PMID 34406128
- [Derived] Katabi LJ, Pu X, Yilmaz HO, Jia Y, Leung S, Duncan AE. Prognostic Utility of KDIGO Urine Output Criteria After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2021 Oct;35(10):2991-3000. doi: 10.1053/j.jvca.2021.02.027. Epub 2021 Feb 13. PMID 33744114
- [Derived] Duncan AE, Jia Y, Soltesz E, Leung S, Yilmaz HO, Mao G, Timur AA, Kottke-Marchant K, Rogers HJ, Ma C, Ince I, Karimi N, Yagar S, Trombetta C, Sessler DI. Effect of 6% hydroxyethyl starch 130/0.4 on kidney and haemostatic function in cardiac surgical patients: a randomised controlled trial. Anaesthesia. 2020 Sep;75(9):1180-1190. doi: 10.1111/anae.14994. Epub 2020 Feb 18. PMID 32072617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 more patients were recruited due to withdrawal (patients did not receive any treatment).
Pre-assignment Details: 9 more patients were recruited to ensure enough power after excluding patients who were randomized but they withdrew from the study and did not receive any treatment (see periods section for details).
Groups:
- HES 130/0.4 (Voluven): 6% HES 130/0.4 during surgery
  HES 130/0.4 (Voluven)
- Human Albumin 5%: human albumin 5% during surgery
  human albumin 5%
Period: Overall Study
Arm/Group | HES 130/0.4 (Voluven) | Human Albumin 5%
Started | 76 | 73
Completed | 69 | 72
Not Completed | 7 | 1
Not completed — Did not receive intervention due to euvolemia | 4 | 1
Not completed — did not receive intervention due to circulatory arrest | 2 | 0
Not completed — did not receive intervention due to logistic reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HES 130/0.4 (Voluven) | Human Albumin 5% | Total
Number analyzed (Participants) | 69 | 72 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (10) | 69 (9) | 70 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 47 | 44 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 62 | 68 | 130
  Not reported | 7 | 4 | 11
Diabetes [Count of Participants; unit: Participants]
  Type 1 | 3 | 0 | 3
  Type 2 | 15 | 20 | 35
Hypertension [Count of Participants; unit: Participants] | 53 | 54 | 107
Stroke [Count of Participants; unit: Participants] | 6 | 3 | 9
Myocardial infarction [Count of Participants; unit: Participants] | 4 | 4 | 8
Surgery type [Count of Participants; unit: Participants]
  Aortic valve only | 35 | 32 | 67
  Aortic valve + CABG | 12 | 16 | 28
  Aortic valve + other | 14 | 18 | 32
  Aortic valve + CABG + other | 8 | 6 | 14
Duration of aortic cross-clamp [Median (Inter-Quartile Range); unit: minutes] | 65 [48 to 91] | 60 [45 to 89] | 62 [46 to 90]
Total fluid [Median (Inter-Quartile Range); unit: L] — total fluid is the amount of colloids and crystalloids during surgery
  L | 2.8 [2.3 to 3.2] | 2.8 [2.1 to 3.7] | 2.8 [2.1 to 3.5]
Transfusion [Count of Participants; unit: Participants] — "Transfusion" Row is reporting the total number of participants who had at least one transfusion
  Participants
    Red blood cell | 13 | 10 | 23
    Platelets | 10 | 10 | 20
    Fresh frozen plasma | 8 | 5 | 13
    Cryoprecipitate | 3 | 4 | 7
    Transfusion | 19 | 16 | 35
Volume of study solution [Median (Inter-Quartile Range); unit: ml] | 500 [400 to 750] | 750 [500 to 1000] | 620 [460 to 800]
Previous cardiac surgery [Count of Participants; unit: Participants] | 13 | 14 | 27
Use of antifibrinolytic drug [Count of Participants; unit: Participants] | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Urine Neutrophil Gelatinase-associated Lipocalin (NGAL) [Time Frame: 24 Hours After Surgery] [Designated as Safety Issue: Yes]
Description: To assess the safety of HES 130/0.4 (Voluven) versus albumin 5% on renal function we will measure urinary concentrations of neutrophil gelatinase-associated lipocalin (NGAL), an important marker of renal function, measured at baseline (following anesthetic induction and prior to surgical incision), at one hour of arrival to intensive care unit (ICU), at 24 hours following completion of surgery.
Time Frame: 3 measurements in total from baseline to 24 hours after surgery: the first one is at baseline; the second one is at one hour of arrive to ICU and last one is at 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | HES 130/0.4 (Voluven) | Human Albumin 5%
Number analyzed (Participants) | 69 | 72
ng/ml
  baseline | 2.9 [1.8 to 5.4] | 4.0 [2.2 to 6.4]
  at 1 hour after surgery | 5.0 [1.4 to 68] | 4.7 [1.6 to 74]
  at 24 hours after surgery | 12 [6.8 to 23] | 15 [7.1 to 22]
Statistical Analysis 1: Comparison: HES 130/0.4 (Voluven) vs Human Albumin 5%; Assuming that NGAL values follow a log normal distribution as in previous studies with a coefficient of variation of 25%, we need 52 patients per group to have 90% power at the 0.025 significance level to be able to claim non-inferiority of HES to albumin using a non-inferiority delta of a ratio of geometric means of 1.15. After Adjusting for the interim monitoring and five potential dropouts and five pilot patients (which were not included in the analyses), we planned to enroll 140 patients; Test type: Non-Inferiority — The non-inferiority delta of a ratio of geometric means is 1.15; p = 0.15, generalized linear model; This analysis used linear mixed model with repeated measurements with an unstructured correlation structure; Geometric mean ratio = 0.91, 95% CI 2-sided [0.57 to 1.44]

2. Secondary Outcome: Kidney Function
Description: Postoperative kidney dysfunction using RIFLE diagnostic criteria was also assessed. Patients were assessed for risk for kidney dysfunction (RIFLE-R), injury to the kidney (RIFLE-I), failure of kidney function (RIFLE-F) using criteria based on only peak serum creatinine concentrations within the first seven postoperative days. Due to too few events, this outcome was redefined to risk (or worse) vs. no risk for this analysis.
  RIFLE classification criteria is listed below:
  Risk (RIFLE-R) Increase in serum creatinine x 1.5 from baseline Injury (RIFLE-I) Increase in serum creatinine x 2 from baseline Failure (RIFLE-F) Increase in serum creatinine x 3 from baseline Loss (RIFLE-L) Complete loss of kidney function > 4 weeks End stage (RIFLE-E) End-stage kidney failure > 3 months
Time Frame: within first 7 postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | HES 130/0.4 (Voluven) | Human Albumin 5%
Number analyzed (Participants) | 69 | 72
Participants
  No risk | 61 | 69
  Risk | 5 | 2
  Injury | 2 | 1
  Failure | 1 | 0
Statistical Analysis 1: Comparison: HES 130/0.4 (Voluven) vs Human Albumin 5%; Test type: Non-Inferiority — the delta for non-inferiority is 1.15; p = 0.92, Chi-squared; Risk Ratio (RR) = 2.78, 95% CI 2-sided [0.64 to 12.1]

3. Secondary Outcome: Postop Urine IL-18
Description: Postop Urine IL-18 (interleukin-18) measured at 1 h of arrival to ICU
Time Frame: postoperative 1 hour
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | HES 130/0.4 (Voluven) | Human Albumin 5%
Number analyzed (Participants) | 69 | 72
pg/ml | 10 [3 to 33] | 16 [5 to 85]
Statistical Analysis 1: Comparison: HES 130/0.4 (Voluven) vs Human Albumin 5%; Test type: Non-Inferiority — the non-inferiority delta was 1.15; p = 0.002, Regression, Linear; IL-18 was log-transformed; geometric mean ratio = 0.45, 5% CI 2-sided [0.21 to 0.95]

4. Secondary Outcome: Postop Urine IL-18
Description: Postoperative urine IL-18 (interleukin-18) measured at 24 hours after surgery
Time Frame: 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | HES 130/0.4 (Voluven) | Human Albumin 5%
Number analyzed (Participants) | 69 | 72
pg/ml | 60 [37 to 91] | 53 [29 to 99]
Statistical Analysis 1: Comparison: HES 130/0.4 (Voluven) vs Human Albumin 5%; Test type: Non-Inferiority — the delta for non-inferiority is 1.15; p = 0.31, Regression, Linear; IL-18 was log-transformed; geometric mean ratio = 0.98, 95% CI 2-sided [0.45 to 2.10]

5. Post Hoc Outcome: Kidney Function
Description: kidney injury using RIFLE criteria based on both peak creatinine levels and urine output, as recommended by Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group
  RIFLE classification criteria is listed below:
  Risk (RIFLE-R) Increase in serum creatinine x 1.5 from baseline urine output < 0.5 mL/kg/hr for more than 6 hrs Injury (RIFLE-I) Increase in serum creatinine x 2 from baseline urine output < 0.5 mL/kg/hr for more than 12 hrs Failure (RIFLE-F) Increase in serum creatinine x 3 from baseline urine output < 0.3 mL/kg/hr for 24 hrs or anuria for 12 hrs Loss (RIFLE-L) Complete loss of kidney function > 4 weeks End stage (RIFLE-E) End-stage kidney failure > 3 months
Time Frame: within the first seven postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | HES 130/0.4 (Voluven) | Human Albumin 5%
Number analyzed (Participants) | 69 | 72
Participants
  No risk | 27 | 16
  Risk | 18 | 24
  Injury | 23 | 31
  Failure | 1 | 0
Statistical Analysis 1: Comparison: HES 130/0.4 (Voluven) vs Human Albumin 5%; Test type: Non-Inferiority — The non-inferiority delta was 1.15; p < 0.001, Chi-squared; Risk Ratio (RR) = 0.8, 95% CI 2-sided [0.61 to 1.03]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HES 130/0.4 (Voluven) | Human Albumin 5%
All-Cause Mortality (participants affected / at risk) | 0/69 | 2/72
Serious Adverse Events (participants affected / at risk) | 17/69 | 12/72
Other Adverse Events (participants affected / at risk) | 0/69 | 0/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HES 130/0.4 (Voluven) (N=69) | Human Albumin 5% (N=72)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
cardiac-related (Cardiac disorders) | 13 (15) | 7 (7)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nervous disorder (Nervous system disorders) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
respiratory related event (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT02192502/Prot_SAP_000.pdf